CLINICAL TRIAL: NCT05161728
Title: Individualisation of Management With Novel Upfront Therapies in Newly Diagnosed Metastasized Prostate Cancer Using (PSMA)PET/CT Imaging
Brief Title: PSMA Response in Metastasized Hormone Sensitive Prostate Cancer
Acronym: PET-MaN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Roderick van den Bergh (Other)
Responsible Party: Sponsor-Investigator, Roderick van den Bergh, Dr. Roderick CN van den Bergh, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL77093.041.21
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: psma; response; metastasis; upfront
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA response evaluation arm (Experimental): PSMA-PET/CT response evaluation, 2 months after starting hormonal therapy, 2 months after starting upfront therapy
  Interventions: Diagnostic Test: PSMA-PET/CT

INTERVENTIONS:
Diagnostic Test: PSMA-PET/CT — PSMA-PET/CT

SUMMARY:
PSMA-PET/CT response measurements after LHRH agonist and upfront therapy in men diagnosed with de novo metastasized hormonal sensitive prostate cancer.

DETAILED DESCRIPTION:
Rationale: Men, newly diagnosed with metastasized prostate cancer on PSMA PET/CT, who start on standard hormonal therapy, are additionally treated with either upfront chemotherapy or upfront extra androgen-receptor targeted agents ('ARTA'), as per guidelines' recommendations. The benefit in overall survival of these two options is similar, but important differences exist in patient-specific efficacy, costs, side-effects, and impact on quality of life. No predictive factors are available to individualize treatment choice. Currently, a one-size-fits-all strategy with hormonal therapy plus chemotherapy is usually followed.

Objective: To assess the predictive value of early response measurements on PSMA-PET/CT for therapy success, defined as time to development of castration-resistant prostate cancer (CRPC), in order to personalize treatment choice.

Study design: Prospective, single arm, open label, non-interventional, non-therapeutic observational cohort study.

Study population: Patients >18 years with newly diagnosed, histologically proven prostate cancer with >3 skeletal or visceral metastatic lesions on the PSMA-PET/CT, who are considered eligible for upfront therapy (apalutamide or abiraterone) in addition to standard hormonal therapy.

Main study parameters/endpoints:

Primary parameter: Predictive value of early response on PSMA-PET/CT to upfront therapy, according to PERCIST criteria. Primary endpoint: Time to development of CRPC. Secondary parameters: Predictive value of early response on PSMA-PET/CT to hormonal therapy; predictive value of baseline PSMA-PET/CT, analysis of response in different subgroups of patients: e.g. high versus low tumour load, high versus low PSA, high versus low Gleason score. Secondary endpoint: Time to initiation of second line therapy after castration-resistant disease has been found.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness:

Patients will be treated according to standard of care, including baseline PSMA-PET/CT. The timing of follow-up PSMA-PET/CT imaging will be standardized. Instead of imaging at biochemical or clinical signs of disease progression, one PSMA-PET/CT will be performed after two months of hormonal therapy, one PSMA-PET/CT will be performed after two months of upfront therapy. Each PSMA-PET/CT scan will require an extra visit (2-3 hours) and a limited radiation burden after intravenous injection of PSMA. The additional information from the standardized follow-up PSMA-PET/CT scans will not be used for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Men >18 years of age.
* Mentally competent and understanding of benefits and potential burden of the study.
* Written and signed informed consent.
* Histological confirmed diagnosis of adenocarcinoma of the prostate.
* Indicated to start on hormonal therapy (any LHRH agonist or antagonist).
* Indicated to start on upfront therapy (apalutamide or abiraterone).
* Any initial PSA.
* Any Gleason score.
* Any T-stage.
* Any N-stage.
* Stage M1, with multiple / high volume metastasis: More than three (>3) metastatic lesions (any combination of either lymph node metastasis outside of pelvis, bone metastasis, or visceral metastasis), as seen on PSMA-PET/CT-imaging. As these patients are treated with palliative intent.

Exclusion Criteria:

* Concomitant malignancy (except from BCC of the skin).
* History of prior diagnosed or treated PCa.
* Any unrelated illness (e.g. active infection, inflammation or laboratory abnormalities) that in the judgment of the investigator will significantly affect patient's clinical status and/or outcome of the study.
* Any known allergy for the upfront therapy.
* Any known allergy for LHRH agonist or antagonist.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2025-10-19 (Estimated); Study Completion 2025-10-19 (Estimated)

PRIMARY OUTCOMES:
CRPC | 18-24 mo after inclusion
  Development of castration-resistant prostate cancer

SECONDARY OUTCOMES:
2nd line therapy | 18-24 mo after inclusion
  Initiation of second line therapy for CRPC

CONTACTS AND LOCATIONS:
Overall Officials: Marnix Lam, MD PhD, Study Chair — UMC Utrecht
Locations (4):
- Netherlands (4):
  - Meander MC, Amersfoort
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - St Antonius Ziekenhuis, Utrecht
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT05161728/Prot_SAP_000.pdf